CLINICAL TRIAL: NCT04611542
Title: Evaluation of Phase I Fathering In Recovery Prototype
Brief Title: Fathering In Recovery
Acronym: FIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DA052949; R43DA052949-01 (NIH)
Record Dates: First submitted 2020-10-28; First posted 2020-11-02 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Parenting; Opioid-use Disorder; Father-Child Relations; Fathers
Keywords: fathers; relapse prevention; opioid-use disorder; behavioral parent training
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FIR Prototype Evaluation (Experimental): 30 fathers in recovery from opioid-use disorder will receive the prototype FIR online intervention.
  Interventions: Behavioral: Fathering In Recovery

INTERVENTIONS:
Behavioral: Fathering In Recovery — Fathering In Recovery (FIR) will be designed to address the unique needs of fathers in treatment for opioid misuse. FIR integrates evidence-based parenting interventions that have well-documented positive outcomes on children, parents, and families, with innovative web-based mobile technology to maximize accessibility, fidelity, and consistency of intervention and support.

SUMMARY:
The majority of men experiencing opioid use disorder and receiving treatment are fathers. Substance use, transitions between in-patient and out-patient treatment, and reunification as a family, all create considerable strain and are predictive of a host of negative long-term outcomes including increased rates of relapse for fathers and elevated risk for behavioral, emotional, and substance use problems in their children. Evidence-based parenting interventions for fathers are lacking in general, yet are exceedingly rare for fathers participating in opioid use disorder treatment, even though the extant research literature suggests the integration of services is not only timely but may help engage and retain fathers in treatment and produce protective factors for children. The goal of this project is to develop and evaluate a prototype of a usable innovative web-based program that integrates existing evidence-based parenting programs, yet tailored specifically to fathers with opioid use disorder and designed for the opioid treatment context in order to promote the implementation and dissemination of father specific empirically-supported treatment.

DETAILED DESCRIPTION:
Investigators will recruit participants for this project through substance use treatment centers in Oregon. Recruitment for the 30 fathers for the evaluation testing will be coordinated in collaboration with substance use treatment center staff members who will contact potentially eligible fathers to give a brief description of the project and ask for permission for Oregon Research Behavioral Intervention Strategies (ORBIS) staff to contact them to provide further information about the study. Fathers that do not give permission for treatment center staff will not be contacted by ORBIS, though they can contact ORBIS directly using the contact information in a brochure that they will receive from treatment centers. Once treatment center staff receive permission from a father for ORBIS to contact them, project staff will call to further explain the details of the project, confirm eligibility requirements and discuss confidentiality. If the father expresses interest in participating, we will send him an information packet and schedule an interview (or a visit if we feel that is necessary to ensure that he understands the project and what we are asking of him).

A total of 30 individual fathers that are eligible and consent to participate will be enrolled in the study. Over a 5-week period (1 week for pretest assessments, 3 weeks for training and skills practice, 1 week for posttest assessments) fathers will participate in using the Fathering In Recovery (FIR) program. To address promise of efficacy, the primary approach for the evaluation of the phase I prototype will be by assessing improvements on pre-intervention to post-intervention outcomes including, parenting knowledge, parenting efficacy, parenting skill, and pre-post reductions in substance use. Fathers will receive a total of $200 for participation in the study.

ELIGIBILITY:
Inclusion:

1. Father with at least part time custody of at least one child between the ages 3-12
2. In recovery from OUD
3. English-speaking
4. Abstinent from substances other than marijuana and alcohol for no more than 1 year
5. Has access to technology allowing for watching internet-based videos such as a smart phone or similar device. Participants will be screened for eligibility criteria by Influents Innovations staff.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Jones, Ph.D., Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD that underlie results in a publication will be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available upon completion of final analysis and publication of results.
Access Criteria: Correspondence via email with the lead author of the publication will be necessary to access to de-identified IPD that underlie results in a publication.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FIR Prototype Evaluation
Started | 30
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention Fathers: Thirty fathers were recruited, consented, and participated in the baseline assessment. Twenty-eight of those fathers engaged in the four-week Fathering in Recovery online intervention and were retained for the post-test (completed one week after program completion - week 5).
Arm/Group | Intervention Fathers
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Parenting Practices Interview
Description: Three sub-scales from the Parenting Practices Interview (PPI): harsh discipline (11 items), inept discipline (9 items), and pro-social parenting. The items are coded on a 7-point scale (1-7) with higher meaning better outcomes. Subscales are averaged to compute a total score.
Time Frame: [Baseline (pretest) & 5 weeks (posttest)] Change in parenting practices from baseline to 5 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fathers Participating in the FIR Program: Twenty-eight fathers that participated in the FIR program and completed the pretest and posttest.
Arm/Group | Fathers Participating in the FIR Program
Number analyzed (Participants) | 28
score on a scale
  Pretest | 2.84 (.70)
  Posttest | 3.83 (.52)
Statistical Analysis 1: Comparison: Fathers Participating in the FIR Program; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 1.02

2. Primary Outcome: Parenting Efficacy
Description: Four 6-item subscales from the Tool for measuring Parent Self-Efficacy (TOPSE): measuring domains of play and enjoyment, discipline practices, perceived control in parenting, and acceptance of parenting role. The items are coded on an 11-point scale (0-10) with higher meaning better outcomes. Subscales are averaged to compute a total score.
Time Frame: [Baseline (pretest) & 5 weeks (posttest)] Change in parenting efficacy from baseline to 5 weeks
Population: Twenty-eight fathers who participate in the FIR intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fathers Changes in Parenting Efficacy: Testing whether the fathers who participated in the FIR program increased their parenting efficacy.
Arm/Group | Fathers Changes in Parenting Efficacy
Number analyzed (Participants) | 28
score on a scale
  Pretest | 6.27 (1.29)
  Posttest | 7.39 (.91)
Statistical Analysis 1: Comparison: Fathers Changes in Parenting Efficacy; Test type: Superiority; p < .001, t-test, 2 sided; Median Difference (Final Values) = 1.12

3. Primary Outcome: Program Knowledge
Description: Knowledge will be assessed to determine the extent to which participants understand basic knowledge delivered in the program. Knowledge items will be derived from conceptual and practical content lessons. 18 items derived from the content on emotion regulation, good directions, and encouragement, will be assessed using multiple-choice questions on a questionnaire developed by the researchers. The items are coded on an 11-point scale (0-10) with higher meaning better outcomes. Subscales are averaged to compute a total score.
Time Frame: [Baseline (pretest) & 5 weeks (posttest)] Change in program knowledge from baseline to 5 weeks
Population: Twenty-eight fathers that engaged in the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Fathers: Thirty fathers engaging in the Fathering In Recovery Online intervention for 4 weeks.
Arm/Group | Intervention Fathers
Number analyzed (Participants) | 28
score on a scale
  Pretest | 2.54 (1.43)
  Posttest | 8.86 (.37)
Statistical Analysis 1: Comparison: Intervention Fathers; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 6.32 — Investigators tested whether pretest to posttest change was significantly greater than 0 at P < 0.05

ADVERSE EVENTS:
Time Frame: 5 weeks.
Arm/Group | FIR Prototype Evaluation
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT04611542/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT04611542/ICF_001.pdf